CLINICAL TRIAL: NCT00307476
Title: A Clinical Comparison of the Rectal Trumpet and Standard Care in Acutely Ill Patients With Fecal Incontinence
Brief Title: Comparison of Rectal Trumpet and Standard Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit target enrollment numbers
Sponsor: Christiana Care Health Services (Other)
Collaborators: American Association of Critical Care Nurses (Other); Wound Ostomy Continence Nurses Society and Hollister (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24200
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Fecal Containment Devices; Skin Integrity
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rectal trumpet (Active Comparator): Patients meeting all study criteria will be randomized to either the rectal trumpet group or the standard treatment.
  For placement of rectal trumpet (Rusch nasopharyngeal airway-32FR):
  Interventions: Device: Rusch Nasopharyngeal Airway
- standard treatment (Other): Patients meeting all study criteria will be randomized to either the rectal trumpet group or the standard treatment. The Numeric Pain Intensity Scale (0-10) or staff observation of physiological indicators (e.g., restlessness, sweating, tachycardia, lacrimation, pupil dilatation, poor ventilator synchrony) for disoriented or unresponsive patients will be used prior to and immediately after placement of either device in order to assess patient comfort. Comfort will be assessed every 8 hours on all oriented patients using the Numeric Pain Intensity Scale.
  Interventions: Device: Rusch Nasopharyngeal Airway

INTERVENTIONS:
Device: Rusch Nasopharyngeal Airway — For placement of rectal trumpet (Rusch nasopharyngeal airway-32FR): Patient's skin is cleansed with Smith and Nephew Personal cleanser and rinsed thoroughly with water to remove any soap residue and dried. Apply 3M no sting barrier film to provide skin protectant. Attach the shaft end of the trumpet to a urinary drainage bag. Using hemostats, clamp the tubing beneath the sample port of the drainage bag. Instill 5cc of mineral oil through the flange end of the trumpet, being careful not to over fill or spill mineral oil onto flange. Release the clamp and allow the mineral oil to drain into urinary drainage bag. If possible, place patient into side-lying position with knees drawn toward the chest. Fold flange into quarters, insert into the rectum. Pull back gently until there is slight resistance. Secure the drainage bag to the bed frame. Drainage tubing should be positioned to prevent tension or pull on trumpet.

SUMMARY:
Primary: To determine the effectiveness of the rectal trumpet compared to the standard care in maintaining skin integrity in patients with fecal incontinence.

Hypothesis (H1): There will be no difference in the failure rates of rectal area skin integrity between subjects receiving the rectal trumpet and those receiving treatment as usual (staqndard care).

Secondary: To determine the ease of use, cost-effectiveness, and level of patient comfort with the rectal trumpet compared to the standard care in patients with fecal incontinence.

Secondary (exploratory) hypotheses:

There will be differences in the ease of use of the devices, costs of the devices, and patient comfort relative to the devices.

DETAILED DESCRIPTION:
Method:

Subjects:

A convenience sample of 80 adult male and female patients in the Wilmington Intensive Care Unit (WICU), Surgical Critical Care Center (SCCC), Medical Intensive Care Unit (MICU), and 6D Step-Down, TSU, 5A, 5E/W, will be recruited. After obtaining informed consent, subjects will be randomized to one of two groups (experimental: rectal trumpet or standard treatment: Hollister fecal incontinent collector).

Inclusion Criteria: Patients who meet the following criteria:

1. Diarrhea - two episodes of loose or watery stool in a 12 hour period
2. ≥ 18 years of age
3. English-speaking patient or guardian
4. Intact skin, may be discolored without breakdown
5. Doctor's order for rectal trumpet (if randomized to treatment group)

Exclusion Criteria: Patients will be excluded from this study if any of the following are present:

1. prolapsed anal sphincter
2. active rectal bleeding
3. colorectal cancer
4. bleeding precautions
5. rectal tone rated 1 (gaping) or 2 (lax)

Instruments:

The data collection instruments used in this study are investigator-developed (see Appendix A - Data Collection Tool). Data will be collected by study and unit nurses at baseline, every eight hours, and PRN throughout the duration of the study. Data will have subject identification removed and subject number assigned.

Digital pictures of patients with any identifying marks (e.g., tattoos, birthmarks, piercings) will have these marks edited out.

Procedure:

A comparison study will be conducted. The staff nurse will identify patients with two or greater episodes of loose or watery stool in a 12 hour period and contact study team. Study team member will determine if patient meets additional inclusion criteria #2, #3, #4, and #5 and does not have exclusion criteria #1, #2 or #3. Once this is determined, the study team member will approach patient or family for consent to participate in study. After consent is obtained, study team member will evaluate patient for remaining exclusion criteria (#4). Rectal tone will be assessed and rated by performing a digital rectal exam. If assessed tone is rated gaping (1) or lax (2), patient is excluded from study.

Patients meeting all study criteria will be randomized to either the rectal trumpet group or the standard treatment. The Numeric Pain Intensity Scale (0-10) or staff observation of physiological indicators (e.g., restlessness, sweating, tachycardia, lacrimation, pupil dilatation, poor ventilator synchrony) for disoriented or unresponsive patients will be used prior to and immediately after placement of either device in order to assess patient comfort. Comfort will be assessed every 8 hours on all oriented patients using the Numeric Pain Intensity Scale.

For placement of rectal trumpet (Rusch nasopharyngeal airway-32FR): Patient's skin is cleansed with Smith and Nephew Personal cleanser and rinsed thoroughly with water to remove any soap residue and dried. Apply 3M no sting barrier film to provide skin protectant. Attach the shaft end of the trumpet to a urinary drainage bag. Using hemostats, clamp the tubing beneath the sample port of the drainage bag. Instill 5cc of mineral oil through the flange end of the trumpet, being careful not to over fill or spill mineral oil onto flange. Release the clamp and allow the mineral oil to drain into urinary drainage bag. If possible, place patient into side-lying position with knees drawn toward the chest. Fold flange into quarters, insert into the rectum. Pull back gently until there is slight resistance. Secure the drainage bag to the bed frame. Drainage tubing should be positioned to prevent tension or pull on trumpet.

Staff will be educated on proper placement of both devices and need for reapplication/reinsertion of either device prior to study initiation. Education will be provided to staff on the following units: SCCC, MICU, 6DSD, and WICU.

Study patients will be assessed every 8 hours and PRN for signs of skin breakdown, stool leakage around devices, dislodgement, or discomfort from devices using the Numeric Pain Intensity Scale for oriented patients. Failure of the fecal incontinent collector will include: leakage within 24 hours of application X 2 attempts at placement, or skin breakdown. Failure of the rectal trumpet will include: leakage X 2 around trumpet with proper positioning within a 24 hour period, skin breakdown, expelling trumpet with continuation of diarrhea X 3 in a 24 hour period, or if the oriented patient, when assessed for discomfort every 8 hours, rates discomfort 2 points above previous rating level of discomfort or requests removal of device due to discomfort.

Selected digital pictures of patients' skin will be taken to establish inter-rater reliability with respect to skin assessment and to provide photographic evidence of skin maintenance, healing, or failure with use of either device. A representative from the Medical Photography department will instruct investigators on digital photographing of patients' skin. Completion of trial will be the return of continence, stool becoming formed, discharge from unit of study, or 14 days whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Diarrhea - two episodes of loose or watery stool in a 12 hour period
2. ≥ 18 years of age
3. English-speaking patient or guardian
4. Intact skin, may be reddened without breakdown
5. Doctor's order for rectal trumpet if patient randomized to treatment group

Exclusion Criteria:

1. prolapsed anal sphincter
2. active rectal bleeding
3. colorectal cancer
4. bleeding precautions
5. rectal tone rated 1 (gaping) or 2 (lax)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2007-06-25 (Actual); Study Completion 2007-06-25 (Actual)

PRIMARY OUTCOMES:
Skin integrity

SECONDARY OUTCOMES:
Ease of use
Cost effectiveness
Patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Denise Netta-Turner, BSN, Principal Investigator — Christiana Care Health Systems
Locations (2):
- United States (2):
  - Christiana Care Health Systems, Newark, Delaware
  - Christiana Care Health Systems-Wilmington, Wilmington, Delaware

IPD SHARING:
Plan to Share IPD: No
inadequate data to share